CLINICAL TRIAL: NCT01241318
Title: Impact of Chlorhexidine Cord Cleansing for Prevention of Neonatal Mortality in Zambia
Brief Title: Zambia Chlorhexidine Application Trial
Acronym: ZamCAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Ministry of Health, Zambia (Other Government); Zambia Center for Applied Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-29647
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-07

CONDITIONS: Sepsis
Keywords: neonate; omphalitis; neonatal mortality; maternal health; umbilical cord infection
MeSH Terms: conditions — Sepsis | interventions — chlorhexidine gluconate; Anti-Infective Agents, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine cord care (Experimental): Mothers located in health facility catchment areas assigned to this arm will apply Chlorhexidine gluconate (4%) to their infants daily until three days after the cord completely separates. Bottles of chlorhexidine is provided to women during antenatal care.
  Interventions: Drug: Chlorhexidine gluconate (4%)
- Dry cord care (Active Comparator): Mothers in health facility catchment areas assigned to this arm will use dry cord care - keeping their babies' umbilical stumps clean and dry - as per normal routine standard of care and in accordance with Zambia Ministry of Health policy.
  Interventions: Procedure: Dry cord care

INTERVENTIONS:
Drug: Chlorhexidine gluconate (4%) — Chlorhexidine is a topical antiseptic that has long been tested for safety and widely used in developed country hospitals, pre-surgical antiseptic technique, wound cleaning and disinfection. Mothers will be instructed to apply 10 ml of 4% chlorhexidine once a day following the infants bath every day from birth until three days after the cord completely separates from the infant's body.
  Other Names: topical antiseptic
  Arms: Chlorhexidine cord care
Procedure: Dry cord care — Mothers will be instructed to keep their infants' umbilical cord stumps clean and dry and to not apply any foreign substances to the cord stump.
  Arms: Dry cord care

SUMMARY:
This will be a cluster-randomized controlled trial to assess whether washing the umbilical cord with a disinfectant (4% chlorhexidine) helps to reduce neonatal deaths in Zambia when compared to the current standard of care, dry cord care.

DETAILED DESCRIPTION:
The primary goals of the Zambia Chlorhexidine Application Trial (ZamCAT) are to assess whether daily 4% chlorhexidine cord cleansing is more effective than dry cord care for the prevention of neonatal deaths and omphalitis (umbilical cord infection) in Southern Province, Zambia. Secondary goals are to 1) compare where pregnant women plan to deliver and where they actually deliver, and 2) to describe the health services network available to pregnant and postpartum women in case of serious illness among the women and their newborn infants.

Clusters consisting of individual health centers and their respective catchment areas will be assigned to one of two arms. In the intervention clusters, mothers will apply 4% chlorhexidine to their infants daily until 3 days after the cord completely separates. Mothers in the control clusters will use dry cord care as per normal routine standard of care and in accordance with Zambia Ministry of Health policy.

In order to achieve the 4th Millennium Development Goal of reducing child mortality by two-thirds, simple, inexpensive, and scalable interventions are required. If the use of a 4% chlorhexidine umbilical cord wash effectively reduces neonatal mortality, this will be a low-cost intervention that can be easily translated from a research project into a program for countrywide implementation in Zambia. These results will also add to the limited evidence base about the effectiveness of interventions for reduction of neonatal mortality in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the 2nd or 3rd trimester
* Age 15 years and above
* Pregnant women who plan to stay in the study area (catchment area of the health facility) for delivery and one month post partum
* Willingness to provide cord care as per the protocol of their cluster
* Willingness to provide informed consent

Exclusion Criteria:

* Pregnant women who are not willing to provide cord care as per the protocol of their cluster
* Pregnant women who are not willing to provide informed consent
* Pregnant women in the 1st trimester
* Pregnant women under age 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women so only women 15 and older
Enrollment: 77535 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davidson H Hamer, MD, Principal Investigator — Boston University Center for Global Health and Development; Katherine Semrau, PhD, Principal Investigator — Boston University Center for Global Health and Development
Locations (1):
- Facilities throughout Southern Province, Choma, Southern Province, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mullany LC, El Arifeen S, Winch PJ, Shah R, Mannan I, Rahman SM, Rahman MR, Darmstadt GL, Ahmed S, Santosham M, Black RE, Baqui AH. Impact of 4.0% chlorhexidine cleansing of the umbilical cord on mortality and omphalitis among newborns of Sylhet, Bangladesh: design of a community-based cluster randomized trial. BMC Pediatr. 2009 Oct 21;9:67. doi: 10.1186/1471-2431-9-67. PMID 19845951
- [Background] Mullany LC, Darmstadt GL, Khatry SK, Katz J, LeClerq SC, Shrestha S, Adhikari R, Tielsch JM. Topical applications of chlorhexidine to the umbilical cord for prevention of omphalitis and neonatal mortality in southern Nepal: a community-based, cluster-randomised trial. Lancet. 2006 Mar 18;367(9514):910-8. doi: 10.1016/S0140-6736(06)68381-5. PMID 16546539
- [Background] Arifeen SE, Mullany LC, Shah R, Mannan I, Rahman SM, Talukder MR, Begum N, Al-Kabir A, Darmstadt GL, Santosham M, Black RE, Baqui AH. The effect of cord cleansing with chlorhexidine on neonatal mortality in rural Bangladesh: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1022-8. doi: 10.1016/S0140-6736(11)61848-5. Epub 2012 Feb 8. PMID 22322124
- [Background] Soofi S, Cousens S, Imdad A, Bhutto N, Ali N, Bhutta ZA. Topical application of chlorhexidine to neonatal umbilical cords for prevention of omphalitis and neonatal mortality in a rural district of Pakistan: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1029-36. doi: 10.1016/S0140-6736(11)61877-1. Epub 2012 Feb 8. PMID 22322126
- [Derived] Solomon H, Henry EG, Herlihy J, Yeboah-Antwi K, Biemba G, Musokotwane K, Bhutta A, Hamer DH, Semrau KEA. Intended versus actual delivery location and factors associated with change in delivery location among pregnant women in Southern Province, Zambia: a prespecified secondary observational analysis of the ZamCAT. BMJ Open. 2022 Mar 7;12(3):e055288. doi: 10.1136/bmjopen-2021-055288. PMID 35256443
- [Derived] Park JH, Hamer DH, Mbewe R, Scott NA, Herlihy JM, Yeboah-Antwi K, Semrau KEA. Components of clean delivery kits and newborn mortality in the Zambia Chlorhexidine Application Trial (ZamCAT): An observational study. PLoS Med. 2021 May 5;18(5):e1003610. doi: 10.1371/journal.pmed.1003610. eCollection 2021 May. PMID 33951036
- [Derived] Henry EG, Semrau K, Hamer DH, Vian T, Nambao M, Mataka K, Scott NA. The influence of quality maternity waiting homes on utilization of facilities for delivery in rural Zambia. Reprod Health. 2017 May 30;14(1):68. doi: 10.1186/s12978-017-0328-z. PMID 28558800
- [Derived] Semrau KEA, Herlihy J, Grogan C, Musokotwane K, Yeboah-Antwi K, Mbewe R, Banda B, Mpamba C, Hamomba F, Pilingana P, Zulu A, Chanda-Kapata P, Biemba G, Thea DM, MacLeod WB, Simon JL, Hamer DH. Effectiveness of 4% chlorhexidine umbilical cord care on neonatal mortality in Southern Province, Zambia (ZamCAT): a cluster-randomised controlled trial. Lancet Glob Health. 2016 Nov;4(11):e827-e836. doi: 10.1016/S2214-109X(16)30215-7. Epub 2016 Sep 29. PMID 27693439
- [Derived] Hamer DH, Herlihy JM, Musokotwane K, Banda B, Mpamba C, Mwangelwa B, Pilingana P, Thea DM, Simon JL, Yeboah-Antwi K, Grogan C, Semrau KE. Engagement of the community, traditional leaders, and public health system in the design and implementation of a large community-based, cluster-randomized trial of umbilical cord care in Zambia. Am J Trop Med Hyg. 2015 Mar;92(3):666-72. doi: 10.4269/ajtmh.14-0218. Epub 2015 Feb 2. PMID 25646254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the 90 clusters (i.e. government-run health facilities), pregnant women who met eligibility criteria attending antenatal care were offered enrollment. Recruitment started February 15, 2011 and ended January 30, 2013.
Pre-assignment Details: Mothers were enrolled in the study while pregnant and infants were enrolled after delivery; thus the total protocol enrollment is women + infants. Study reporting is completed at the woman level and thus the total enrolled is listed at the woman level in the outcomes tables.
Groups:
- Chlorhexidine Cord Care: Mothers located in health facility catchment areas assigned to this arm will apply chlorhexidine to their infants daily until three days after the cord completely separates.
  Chlorhexidine gluconate (4%): Chlorhexidine is a topical antiseptic that has long been tested for safety and widely used in developed country hospitals, pre-surgical antiseptic technique, wound cleaning and disinfection. Mothers will be instructed to apply 10 ml of 4% chlorhexidine once a day following the infants bath every day from birth until three days after the cord completely separates from the infant's body.
Period: Overall Study
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care
Started | 19629 (Women enrolled) | 20050 (Women enrolled)
Liveborn Infant | 18510 (Infants) | 19346 (Infants)
Completed | 18450 (Infants) | 19308 (Infants)
Not Completed | 1179 | 742
Not completed — Woman: false pregnancies | 27 | 15
Not completed — Woman: miscarriage/abortion | 46 | 38
Not completed — Withdrawal by Subject | 175 | 46
Not completed — Lost to Follow-up | 740 | 455
Not completed — Death | 2 | 4
Not completed — Withdrew/Lost to Follow after delivery | 60 | 38
Not completed — Woman: Stillborn infant | 129 | 146

BASELINE CHARACTERISTICS:
Population: Pregnant women attending health facilities for antenatal care
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care | Total
Number analyzed (Participants) | 19629 | 20050 | 39679
Age, Customized [Number; unit: participants]
  <20 years | 4671 | 4580 | 9251
  20-35 years | 12772 | 13122 | 25894
  >35 years | 2012 | 2194 | 4206
  Missing (not recorded) | 174 | 154 | 328
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19629 | 20050 | 39679
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Tonga | 17003 | 17650 | 34653
  Ila | 105 | 121 | 226
  Lozi | 786 | 795 | 1581
  Nyanja | 525 | 432 | 957
  Bemba | 413 | 433 | 846
  Other | 629 | 481 | 1110
  Missing (not recorded) | 168 | 138 | 306
Region of Enrollment [Number; unit: participants]
  Zambia | 19629 | 20050 | 39679
Maternal Education [Number; unit: participants]
  No eduction | 1936 | 1958 | 3894
  Lower Primary | 2293 | 2563 | 4856
  Upper Primary | 7731 | 7874 | 15605
  Junior Secondary | 5422 | 5499 | 10921
  Upper Secondary | 1895 | 1840 | 3735
  >Upper Secondary | 180 | 160 | 340
  Do not know | 3 | 10 | 13
  Missing (not recorded) | 169 | 146 | 315
Marital Status [Number; unit: participants]
  Single | 3021 | 3133 | 6154
  Married | 16107 | 16499 | 32606
  Separated, divorced or widowed | 224 | 187 | 411
  Cohabiting | 109 | 89 | 198
  Missing (not recorded) | 168 | 142 | 310
Maternal literacy [Number; unit: participants]
  Not at all | 5037 | 5491 | 10528
  A bit | 8835 | 9516 | 18351
  Very well | 5492 | 4835 | 10327
  No response from mother | 77 | 61 | 138
  Missing (not recorded) | 188 | 147 | 335
Household water source [Number; unit: participants]
  Household tap | 1861 | 1715 | 3576
  Community tap | 1919 | 1761 | 3680
  Other water source on own property | 2295 | 2403 | 4698
  Community well or river | 13241 | 13768 | 27009
  No answer from Mother | 56 | 62 | 118
  Other | 67 | 166 | 233
  Missing (Not recorded) | 190 | 175 | 365
Parity [Mean (Standard Deviation); unit: pregnancies] | 2.4 (2.3) | 2.5 (2.4) | 2.5 (2.4)
Gravida [Mean (Standard Deviation); unit: deliveries] | 3.5 (2.3) | 3.6 (2.4) | 3.6 (2.4)
Gestational Age at enrollment [Mean (Standard Deviation); unit: weeks] | 28.0 (7.2) | 28.4 (7.2) | 28.3 (7.2)
Slept under mosquito bednet the previous night [Number; unit: participants]
  Yes | 11092 | 11783 | 22875
  No | 8310 | 8075 | 16385
  Missing (not recorded) | 227 | 192 | 419

OUTCOME MEASURES:

1. Primary Outcome: All-cause Neonatal Mortality
Description: All-cause neonatal mortality based on vital status at 28 days post-partum
Time Frame: 28 days post-partum
Measure: Number; unit: participants
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care
Number analyzed (Participants) | 18450 | 19308
participants
  Neonatal mortality | 282 | 263
  Survived to day 28 | 18168 | 19045
Statistical Analysis 1: Comparison: Chlorhexidine Cord Care vs Dry Cord Care; Test type: Superiority or Other; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.88 to 1.44] — The chlorhexidine arm is the numerator and dry cord care arm is the denominator in the relative risk calculation. Generalised estimating equation models were used to adjust for cluster randomized design

2. Primary Outcome: All-cause Neonatal Mortality Among Newborns Who Survived at Least First Day of Life
Description: All-cause mortality by day 28 of life among newborns who survive at least the first day of life
Time Frame: 28 days post-partum
Population: All liveborn neonates who survived the first 24 hours after delivery
Measure: Number; unit: neonates who survived first 24 hours
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care
Number analyzed (Participants) | 18424 | 19266
neonates who survived first 24 hours
  Neonatal mortality | 200 | 186
  Survived to day 28 | 18224 | 19080
Statistical Analysis 1: Comparison: Chlorhexidine Cord Care vs Dry Cord Care; Test type: Superiority or Other; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.86 to 1.47] — Generalized estimating equation models adjusting for cluster-randomized design were used

3. Secondary Outcome: Incidence of Omphalitis
Description: Omphalitis, or umbilical cord infection, defined as:
  * presence of umbilical cord pus and mild, moderate or severe redness
  * moderate or severe redness without the presence of umbilical cord pus
Time Frame: 28 days postpartum
Measure: Number; unit: neonates
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care
Number analyzed (Participants) | 18510 | 19346
neonates
  Omphalitis | 82 | 118
  No omphalitis | 18428 | 19228
Statistical Analysis 1: Comparison: Chlorhexidine Cord Care vs Dry Cord Care; Test type: Superiority or Other; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.47 to 1.13] — Generalized estimating equation models adjusting for cluster-randomized design were used

4. Secondary Outcome: Place of Delivery
Description: The location where mothers gave birth (home versus a health facility) will be compared to their planned delivery location.
Time Frame: 28 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care
Number analyzed (Participants) | 18510 | 19346
Participants
  Home Delivery | 6509 | 6682
  Facility Delivery | 11456 | 12204
  Other | 190 | 128
  Missing | 355 | 332

5. Secondary Outcome: Factors Influencing Delivery Location
Description: Health facility characteristics and maternal decision making factors that influence choice of delivery location (health facility vs. home delivery)
Time Frame: 28 days postpartum
Population: Women enrolled in the ZamCAT study and delivery location known. Please note these are different denominators reported as this analysis is not based on intervention randomization, but rather an analysis focused on women's location of childbirth. Therefore, the number of women included in this analysis is based on a subset of all women enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Facility Delivery: Women who enrolled in ZamCAT study and delivered at a facility
- Home Delivery: Women who enrolled in ZamCAT study and delivered at home
Arm/Group | Facility Delivery | Home Delivery
Number analyzed (Participants) | 23815 | 13255
Participants
  Same Location as Prior Delivery | 3198 | 2082
  Need for Skilled Attendance12991 | 12991 | 5693
  Financial Constraints | 1823 | 1249
  Physical Distance | 6345 | 3930
  Relationship with Provider | 572 | 429
  Family/Social Expectations | 1255 | 990
  Safety for Mother/Baby | 14129 | 5911
  Other | 1480 | 803
  Missing | 1364 | 770

6. Secondary Outcome: Health Facility Characteristics
Description: Characterization of the health services available to pregnant women, postpartum women and their offspring as assessed by comprehensive health facility and health worker surveys. This data was assessed and reported on 100 facilities (10 district hospitals and 90 health facilities).
Time Frame: 12 months after study initiation
Population: Health facilities
Measure: Number; unit: Health facilities
Units Other Than Participants: Health facilities
Groups:
- Study Health Facilities & Hospitals: 90 health facilities and 10 district hospitals were included in the main chlorhexidine trial. A survey was completed to assess availability of emergency obstetric care.
Arm/Group | Study Health Facilities & Hospitals
Number analyzed (Participants) | 39679
Number analyzed (Health facilities) | 100
Health facilities
  Basic emergency obstetrical and newborn care | 6
  No basic emergency obstetrical and newborn care | 94

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 1 month follow up period past delivery.
Description: Umbilical cord was observed by the field data collector at every visit (day 1, 4, 10, 28 post-partum). Adverse events were defined as ocular exposure to chlorhexidine, local skin irritation, accidental ingestion, contact dermatitis, or anaphylaxis.
Arm/Group | Chlorhexidine Cord Care | Dry Cord Care
All-Cause Mortality (participants affected / at risk) | 282/18510 | 263/19346
Serious Adverse Events (participants affected / at risk) | 0/18510 | 0/19346
Other Adverse Events (participants affected / at risk) | 9/18510 | 0/19346
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine Cord Care (N=18510) | Dry Cord Care (N=19346)
Chlorhexidine-related adverse events (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
Chlorhexidine ocular exposure (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Only 89% (37 856 of 42 570) of the target sample size was attained. When we completed a post-hoc power calculation with the obtained sample size and observed Neonatal Mortality Rate (NMR), we had 80% power to detect a 28% reduction in NMR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less